CLINICAL TRIAL: NCT00332657
Title: Anecortave Acetate Risk Reduction Trial (AART)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C-05-34
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2009-09

CONDITIONS: AMD
MeSH Terms: interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Anecortave Acetate, 15 mg (Experimental): One 0.5 mL injection of 30 mg/mL Anecortave Acetate Sterile Suspension into the posterior juxtascleral depot (PJD) at 6-month intervals for 42 months.
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL
- Anecortave Acetate, 30 mg (Experimental): One 0.5 mL injection of 60 mg/mL Anecortave Acetate Sterile Suspension into the posterior juxtascleral depot (PJD) at 6-month intervals for 42 months.
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL
- Anecortave Acetate Vehicle (Sham Comparator): One sham injection at 6-month intervals for 42 months. Syringe and vehicle were not inserted into the eye.
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL — One 0.5 mL injection into the PJD at 6-month intervals for 42 months
  Arms: Anecortave Acetate, 15 mg
Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL — One 0.5 mL injection into the PJD at 6-month intervals for 42 months
  Arms: Anecortave Acetate, 30 mg
Other: Anecortave Acetate Vehicle — One 0.5 mL sham injection at 6-month intervals for 42 months. Syringe and vehicle were not inserted into the eye.
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of this study is to demonstrate that Anecortave Acetate for Depot Suspension (15 mg or 30 mg) is safe and effective in arresting the progression of dry age-related macular degeneration (AMD) in patients who are at-risk for progressing to wet AMD.

ELIGIBILITY:
Inclusion Criteria:

* Dry AMD in study eye, Wet AMD non-study eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 50.
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sight-threatening choroidal neovascularization (CNV) in study eye | Month 48

SECONDARY OUTCOMES:
Time to development of sight-threatening CNV | Timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Terry Wiernas, PhD, Study Director — Study Director
Locations (1):
- India, Bangalore, India